CLINICAL TRIAL: NCT04297605
Title: A Pilot Study of Pembrolizumab and Single Agent Chemotherapy as First Line Treatment for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer With Eastern Cooperative Oncology Group (ECOG) Performance Status of 2
Brief Title: Study of Pembrolizumab and Single Agent Chemotherapy as First Line Treatment for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer With Eastern Cooperative Oncology Group (ECOG) Performance Status of 2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Megan Baumgart, Assistant Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULUN19148
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Eastern Cooperative Oncology Group (ECOG); Non-small Cell Lung Cancer; pembrolizumab; performance status of 2 (PS2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Drug Therapy; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental 1: pembrolizumab and Pemetrexed (Experimental): Treatment includes administration of pembrolizumab and chemotherapy, which are administered every 21 days
  Pembrolizumab 200 mg and Pemetrexed 500 mg/m2 day 1 of 21 day cycle (for non-squamous only)
  Interventions: Drug: Pembrolizumab; Other: Pemetrexed (Chemotherapy)
- Experimental 2: pembrolizumab and Nab-paclitaxel (Experimental): Treatment includes administration of pembrolizumab and chemotherapy, which are administered every 21 days
  Pembrolizumab 200 mg and Nab-paclitaxel 100 mg/m2 days 1,8 of 21 day cycle x 4 cycles followed by pembrolizumab alone
  Interventions: Drug: Pembrolizumab; Other: Nab-paclitaxel (Chemotherapy)

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg
Other: Pemetrexed (Chemotherapy) — 500 mg/m2 day 1 of 21 day cycle (for non-squamous only)
  Arms: Experimental 1: pembrolizumab and Pemetrexed
Other: Nab-paclitaxel (Chemotherapy) — 100 mg/m2 days 1,8 of 21 day cycle x 4 cycles
  Arms: Experimental 2: pembrolizumab and Nab-paclitaxel

SUMMARY:
The purpose of this study is to understand if treatment with one chemotherapy medication combined with immune therapy (pembrolizumab) is tolerable and effective for patients with lung cancer and performance status of 2 (PS2), which means you have limitations in carrying out certain activities or spend up to half of your day resting.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be >18 years old at time of diagnosis
2. Histologically confirmed non-small cell lung cancer
3. ECOG PS 2
4. Clinical staging of IIIc or IV disease.

4A. For patients with stage IIIc disease, patients are ineligible for or refuse standard treatment with platinum-double chemotherapy and radiation.

4B. For patients with stage IV disease, platinum doublet chemotherapy is not appropriate, deemed unsafe by the treating physician, or declined by the patient

4C. Screening lab work must meet the following parameters:

4Ca. Absolute neutrophil count (ANC) ≥1000/mm3

4Cb. Platelet count ≥100,000/mm3

4Cc. CrCl>50 (if pemetrexed is to be offered)

4Cd. AST and ALT ≤ 2.5 x ULN

4D. Patients with small, asymptomatic brain metastases are eligible

4E. Women of childbearing potential must be negative for pregnancy testing (urine or blood) and agree to use effective contraception. Viable contraception should be used after trial screening, before initiation of chemotherapy, and throughout the duration of active treatment in the study.

Non-childbearing potential is defined as (by other than medical reasons): -Amenorrheic >2 years

* Amenorrheic for <2 years and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
* Post hysterectomy, oophorectomy or tubal ligation. Otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study drug

  4F.Participants must read or be read and explained the purposes of the study and sign a statement of informed consent prior to participation. Those who do not read or understand English are eligible and may be consented according to institutional regulations.

Exclusion Criteria:

1. Patients with history of autoimmune conditions with the following exceptions, which are allowed: alopecia, vitiligo, rheumatoid arthritis, psoriasis/psoriatic arthritis, Hashimoto's thyroiditis
2. Patients on immunosuppressive medication, including steroids (if doses exceed equivalent of prednisone 10 mg daily). Short courses of steroids which are discontinued prior to start of treatment are acceptable.
3. Patients with cardiovascular, hepatic, or renal systemic diseases that would preclude use of chemotherapy and/or immunotherapy per the treating investigator.
4. The patient must not be on any clinical trials involving other experimental therapies during study treatment
5. Women who are currently pregnant or breast-feeding
6. Patients with any other concurrent medical or psychiatric condition that were deemed inappropriate for entry into the study per the investigator.
7. Symptomatic, untreated brain metastases. Patients with treated brain metastases may be considered eligible after completion of radiation if steroids have been tapered to less than equivalent of 10 mg of prednisone.
8. Active infection requiring IV antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | 18 Months
  Determine the rate of treatment-limiting toxicities in patients with advanced non-small cell lung cancer with ECOG PS 2 who are treated with pembrolizumab and single-agent chemotherapy

SECONDARY OUTCOMES:
Percentage of participants with Complete Response or Partial Response | 18 Months
  Determine the proportion of patients who achieve a complete or partial response as their best overall response based on RECIST v1.1 criteria will be evaluated. Patients with nonevaluable or unknown response status will be considered nonresponders.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Baumgart, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided